CLINICAL TRIAL: NCT05570422
Title: A Phase 1/2 Study to Evaluate the Safety, Tolerability, Preliminary Efficacy of KRC-01 Intratumoral Injection Combined With Radiotherapy in Patients With Locally Advanced Cervical Cancer
Brief Title: A Study to Evaluate the Safety, Tolerability, Preliminary Efficacy of KRC-01
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Kortuc, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: KRC-01-C01
Record Dates: First submitted 2022-08-29; First posted 2022-10-06 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Cisplatin; Drug Therapy; Brachytherapy

STUDY DESIGN:
Intervention Model Description: Phase 1 open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- dose-escalation single arm (Experimental): Dose-escalation single arm, open label study. All eligible subjects will receive external beam radiotherapy (EBRT) with cisplatin (40 mg/m2) intravenously (IV) once weekly for 5 weeks (sixth dose optional) followed by image-guided brachytherapy (BT).
  KRC-01 will be dosed intratumorally within 2 hours prior to EBRT starting from second week of EBRT.
  There are two cohorts (n=5 per cohort) Cohort 1: Once-a-week between Monday to Thursday (not necessarily the same day every week) Cohort 2: Twice-a-week with a 1- or 2- day interval (either Mon+Wed, Mon+Thu, or Tue+Thu)
  Interventions: Drug: KRC-01; Radiation: External Beam Radiation Therapy; Drug: cisplatin; Radiation: brachytherapy

INTERVENTIONS:
Drug: KRC-01 — KRC-01 is a solution that contains hydrogen peroxide 3% with sodium hyaluronate 1%. Hydrogen peroxide is the active ingredient for this radiosensitizer.
Radiation: External Beam Radiation Therapy — * Target definition for EBRT will be based on 3D imaging by computed tomography, positron emission tomography with computed tomography, or MRI.
  * Intensity-modulated radiotherapy (IMRT) must be used.
  * IMRT should be given once daily Monday-Friday, 5 fractions per week.
Drug: cisplatin — * Weekly concomitant cisplatin (40 mg/m2) during EBRT
  * Neo-adjuvant chemotherapy or other forms of antineoplastic treatment apart from weekly concomitant cisplatin (40 mg/m2) are not allowed.
  * Adjuvant chemotherapy (after completion of EBRT+BT) is not allowed.
  Other Names: Chemotherapy
Radiation: brachytherapy — * BT treatment planning will be based on 3D-image-guided BT by MRI.
  * Low-dose-rate, pulsed-dose-rate, or high-dose-rate BT

SUMMARY:
This is a seamless Phase 1/2 study consisting of two components. Phase 1 component is a dose-escalation, single arm, open label study in 10 patients to evaluate the safety and tolerability of KRC 01. Phase 2 component is a randomized, open label, controlled, multi-center study in 60 patients to evaluate the preliminary antitumor effect of KRC-01 in combination with CRT.

DETAILED DESCRIPTION:
This is a seamless Phase 1/2 study consisting of two components. Phase 1 component is a dose-escalation, single arm, open label study in 10 patients to evaluate the safety and tolerability of KRC 01. Phase 2 component is a randomized, open label, controlled, multi-center study in 60 patients to evaluate the preliminary antitumor effect of KRC-01 in combination with CRT.

Phase 1 component (n=10) Phase 1 component is a dose-escalation single arm, open label study. All eligible subjects will receive external beam radiotherapy (EBRT) with cisplatin (40 mg/m2) intravenously (IV) once weekly for 5 weeks (sixth dose optional) followed by image-guided brachytherapy (BT).

KRC-01 will be dosed intratumorally within 2 hours prior to EBRT starting from second week of EBRT.

There are two cohorts (n=5 per cohort) Cohort 1: Once-a-week between Monday to Thursday (not necessarily the same day every week) Cohort 2: Twice-a-week with a 1- or 2- day interval (either Mon+Wed, Mon+Thu, or Tue+Thu)

After 5 subjects of Cohort 1 have completed CRT+BT, the safety review committee (SRC) will evaluate the safety and tolerability of KRC-01 once-a-week dosing and determine Go/ No Go decision to Cohort 2 (twice-a-week dosing).

After all 10 subjects have completed CRT+BT, the SRC will evaluate the safety and tolerability of KRC 01 and determine Go/ No Go decision to Phase 2 component with optimal dosing regimen.

Phase 2 component (n=60) Phase 2 component is a randomized, open label study. All eligible subjects will be randomized to Standard of care (SOC) group or SOC with KRC-01 group.

All subjects will receive EBRT with cisplatin (40 mg/m2) IV once-a-week for 5 weeks (sixth dose optional) followed by image-guided BT. Only for KRC-01 group, KRC-01 will be dosed intratumorally at the optimal dosing schedule selected in Phase 1 component within 2 hours prior to EBRT starting from second week of EBRT.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent before participation.
* Female subjects age 18 years or older.
* Histologically diagnosed squamous cell carcinoma, adenocarcinoma or adeno-squamous cell carcinoma of the uterine cervix.
* FIGO stage II and III locally advanced cervical cancer.
* No evidence of metastatic disease.
* At least one tumor that qualifies as a Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 tumor with tumor size >5 cm diameter, not previously irradiated, at baseline assessed [by magnetic resonance imaging (MRI)] within 28 days before Day 1.
* No prior chemotherapy or radiotherapy for cervical cancer.
* Intention to undergo treatment including EBRT with 5 cycles of cisplatin followed by BT; to be completed within 8 weeks of its initiation.
* Patients with predicted life expectancy of 3 months or more.
* Target tumor is accessible for intratumoral injection.
* Eastern Cooperative Oncology Group (ECOG) Performance status of 0 or 1.
* Negative pregnancy test before start of CRT in women of childbearing potential and an ability/willingness to protect against pregnancy from consent and for 3 months post-RT.

Exclusion Criteria:

* Other primary malignancies except basal cell carcinoma of the skin.
* Histologically diagnosed small cell (neuroendocrine), melanoma, clear cell and other rare variants of the classical adenocarcinoma at cervices.
* Previous pelvic or abdominal radiotherapy.
* Previous total or partial hysterectomy.
* Combination of preoperative radiotherapy with surgery.
* Patients receiving neo-adjuvant chemotherapy or non-protocol antineoplastic treatment apart from weekly cisplatin (40 mg/m2).
* Anatomical location and/or extent of disease difficult to access for safe intratumoral drug injections.
* Contraindications to the pelvic radiation such as inflammatory bowel disease and collagen vascular disease.
* Contraindications to MRI.
* Patients on anticoagulants or deranged coagulation profile.
* Pregnancy or nursing.
* High medical risks because of non-malignant systemic disease or with active uncontrolled infection.
* Participation in another clinical trial with an investigational drug, device or biologic within the preceding 3 months, except an observational study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — females at birth currently with a cervix
Enrollment: 70 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-01-30 (Estimated); Study Completion 2027-03-30 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | 36 month
  An AE is any untoward medical occurrence in a patient or clinical investigation subject administered a study drug that does not necessarily have a causal relationship with the treatment.
AEs of special interest | 36 month
  (local pain, radiation dermatitis, tumor lysis syndrome, superficial soft tissue fibrosis, vaginal stenosis, gastrointestinal/urinary AEs, and severe and medically significant bleeding (requires urgent intervention) after intratumoral injection)
Physical examination | at the time of Screening and at Week 6 and partial examination will be done weekly in between to document relevant changes.
  The physical examination will include:
  * General appearance
  * Head, eyes, ears, nose, and throat
  * Respiratory
  * Cardiovascular
  * Musculoskeletal
  * Abdomen
  * Neurologic
  * Extremities
  * Dermatologic
  * Lymphatic Partial examination, patient will verbally report changes since last week.
Tolerance | week 1 to 6
  • Number of patients who have a significant treatment delays/interruption (total duration > 59 days)

SECONDARY OUTCOMES:
Progression-free survival | : minimum 2 years, maximum 3 years
  PFS is defined as the time from randomization to the first documented PD or death due to any cause, whichever occurs first. Per RECIST 1.1, or by histopathologic confirmation of suspected disease progression, PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions is also considered PD. Unequivocal progression of non-target lesions is also considered PD.
Overall survival | minimum 2 years, maximum 3 years
  mortality rates
Disease-free survival | minimum 2 years, maximum 3 years
  Disease progression can be considered as a worsening of a patient's condition attributable to the disease for which the investigational product is being studied. It may be an increase in the severity of the disease under study and/or increases in the symptoms of the disease. An event can be attributed to disease progression even without radiological or biomarker evidence of disease progression.
  Deterioration of the disease under study and associated symptoms or findings, including the development of new, or the progression of existing, metastases, should not be regarded as an AE, unless the study medication is considered to have contributed to the progression.
Health-related quality of life (QOL) | minimum 2 years, maximum 3 years
  European Organisation for Research and Treatment of Cancer (EORTC) QOL 30-Item Questionnaire (QLQ-C30) and EORTC 24-Item Cervical Cancer Questionnaire (QLQ-CX24)

OTHER OUTCOMES:
CRT poor responder rate | Out to Week 4 or 5
  Poor responder is defined as 40 cc residual tumor at Week 4 or Week 5 assessed by MRI T2) in patients who have > 40cc tumor at the baseline
Feasibility of hypoxia imaging | Screening and after the completion of KRC-01 dosing (between Week 6 to Month 3).
  Diffusion-weighted imaging-MRI (DWI-MRI) and Dynamic contrast-enhanced MRI (DCE-MRI)

CONTACTS AND LOCATIONS:
Locations (5):
- India (2):
  - Site 2, Chandigarh
  - Site 1, Visakhapatnam
- Thailand (2):
  - Site 5, Bangkok
  - Site 4, Chiang Mai
- Site 3, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
undecided